## **HD-OLDER** — Statistical Analysis Plan (SAP)

| Study title: | HemoDiafiltration versus HemoDialysis in OLDER people: a randomized, multicenter, crossover, pragmatic clinical trial |
|---|---|
| Short title / Acronym: | HD-OLDER |
| SAP version/date: | v1.0 — 02-Sep-2025 |
| Protocol reference: | HD-OLDER, Protocol v3 (17-Jul-2025) |
| Sponsor: | Fondation AUB SANTÉ |
| Principal Investigator: | Dr Mabel AOUN |

## 1. Background and rationale

Hemodiafiltration (HDF) and high-flux hemodialysis (HD) are standard dialysis modalities. Very elderly patients (≥85 years) are under-represented in prior trials, and Dialysis Recovery Time (DRT) is a practical, patient-centred endpoint for tolerability. HD-OLDER uses a two-period crossover (HDF↔HD) to enable precise within-patient comparisons in a small, frail population. A two-week low-flux HD washout is implemented at study start and between periods to limit carryover. Pragmatic conduct preserves usual-care practices and enhances external validity.

## 2. Objectives and estimand

## 2.1 Primary objective

To compare the within-period change in DRT (minutes) between HDF and high-flux HD over each 3-month period.

#### 2.2 Secondary objectives

To compare, between modalities, changes in: fatigue (SONG-Fatigue 0–9), functional performance (STS-30), health-related quality of life (SF-12 PCS/MCS); and counts per period of symptomatic intradialytic hypotension and circuit clotting; changes in laboratory markers and dialysis adequacy (Kt/V); and safety (deaths, hospitalizations).

#### 2.3 Estimand (primary)

- **Population:** All randomized patients ≥85 years who enter the treatment periods.
- Variable: Period-level change in DRT: mean(end-of-period window) mean(start-of-period window), minutes.
- Intercurrent events: Treatment-policy strategy (analyse as randomized regardless of adherence, hospitalizations, etc.).
- **Summary measure:** Adjusted mean difference (HDF HD) from a linear mixed-effects model (LMM) with fixed effects for modality, period, sequence, centre; random intercept for patient; and pre-specified covariates.
- **Population-level interpretation:** Average causal effect of allocating HDF vs HD on within-period change in DRT, in the intended pragmatic setting.

## 3. Hypothesis framework and error control

Confirmatory framework: Superiority for the primary endpoint only. Null (H0): Mean change in DRT is the same under HDF and HD ( $\beta_1 = 0$ ).

Alternative (H1): HDF reduces DRT ( $\beta_1 < 0$ ).

**Type I error:** Two-sided  $\alpha = 0.05$ ; report 95% Cls.

Multiplicity: None for secondaries (estimation-focused with 95% CIs and two-sided

p-values, descriptive interpretation). No hierarchical testing.

## 4. Study design overview

- Design: Randomized (1:1) two-sequence, two-period crossover; sequences A (HDF→HD) and B (HD→HDF).
- Periods: Each 3 months.
- Washout: Two weeks of low-flux HD at study start and between periods.
- **Blinding:** Not feasible for patients/clinicians; statisticians analyse anonymised treatment codes where possible.
- **Centres:** Ten dialysis units in France.

• **Planned sample size:** 62 randomized (targeting ≥56 evaluable).

## 5. Analysis populations

- Intention-to-treat (ITT) primary: All randomized, analysed as randomized and per period modality, irrespective of adherence or deviations.
- Per-protocol (PP) sensitivity: ITT subset completing both periods; ≥80% of attended sessions on allocated modality in each period; valid start and end windows for the endpoint in the period; exclude major deviations (e.g., inadequate washout, cross-over contamination).
- Safety set: All randomized with ≥1 post-randomization dialysis session; safety attributed to modality received within each period (as-treated by session aggregation).

#### 6. Outcomes and derivations

#### 6.1 Primary endpoint — DRT (minutes)

- Question: "How long did it take you to recover from your last dialysis session?"
- **Schedule:** Start (~week 0), Mid (~6 weeks), End (~12 weeks) in each period. At each window, obtain up to three consecutive sessions.
- Window rule: Compute the window mean if ≥2 of 3 session values are available; otherwise the window is missing.
- **Derivation:** Period-level change = mean(End) mean(Start). Negative values indicate faster recovery (improvement).

## 6.2 Secondary endpoints

- **SONG-Fatigue (0–9):** Sum of three items (all required). Change = End Start per period.
- **STS-30:** Mean repetitions over three consecutive sessions per window; Change = End Start.
- **SF-12 PCS/MCS:** Baseline and End of each period; Change = End Start.
- **Counts per period:** Total symptomatic intradialytic hypotension; total circuit clotting.
- **Laboratories & adequacy:** Haemoglobin, albumin, potassium, phosphate, Kt/V as priority; other routine labs exploratory. Change = month 3 baseline month.
- Safety: Deaths and hospitalizations per period; exposure-adjusted incidence rates.

## 7. Sample size and information size

• **Planned N:** 62 randomized, anticipating ≥56 evaluable.

**Justification:** Prior data in  $\geq$ 85-year-olds indicate large between-modality differences in mean DRT with wide SDs. The current N achieves  $\approx$ 80% power (two-sided  $\alpha$ =0.05) under conservative parallel-group assumptions. The crossover design is expected to yield greater precision than this conservative calculation by exploiting within-patient comparisons. No interim analysis or re-estimation is planned.

## 8. General analysis conventions

- **Data cut:** Final database lock after Period-2 ends for the last participant and all queries are resolved.
- Units: DRT in minutes (convert hours to minutes).
- **Transformations:** Primary on the minute scale for interpretability; log[DRT+1] sensitivity if residual skewness persists.
- **Rounding:** Descriptives to one decimal where appropriate; effect estimates to one decimal (minutes) and 2–3 significant figures for ratios.
- Covariates (pre-specified): Age, sex, dialysis vintage, access type (AVF/AVG vs CVC), baseline DRT at period start.

## 9. Primary analysis

#### 9.1 Model

Unit of analysis: patient-period.

For patient *i* in period p (p=1,2):

Change\_ $\{i,p\} = \beta_0 + \beta_1 \cdot Modality_{\{i,p\}} + \beta_2 \cdot Period2_{\{p\}} + \beta_3 \cdot Sequence_{\{i\}} + \beta_4 \cdot Centre_{\{i\}} + X'_{\{i,p\}}\gamma + u_{\{i\}} + \epsilon_{\{i,p\}},$ 

with  $u_{i} \sim N(0, \tau^{2})$  (random intercept),  $\varepsilon_{i} \sim N(0, \sigma^{2})$ .

- Modality: 1 = HDF, 0 = high-flux HD.
- Period2: 1 if period 2, else 0.
- Sequence: 1 = HDF→HD, 0 = HD→HDF.
- Centre: fixed categorical effect.
- X: pre-specified covariates listed in §8.

**Target parameter:**  $\beta_1$  = adjusted mean difference in within-period DRT change (HDF – HD), minutes;  $\beta_1$  < 0 favours HDF.

**Estimation:** REML. Report  $\beta_1$  with 95% CI and two-sided p-value.

#### 9.2 Decision rule

Conclude HDF superiority if  $\beta_1$  < 0 and the 95% CI excludes 0. Otherwise, no superiority is concluded.

#### 9.3 Carryover assessment and fallback

- Definition: Residual influence of Period-1 modality on Period-2 outcomes despite washout.
- Screen: Test Modality × Period interaction (diagnostic threshold p<0.10).
- Fallback if flagged: Primary inference switches to Period-1-only ITT
  parallel-groups ANCOVA of Period-1 change (factors: modality, sequence;
  covariate: baseline DRT at Period-1 start). Provide Wilcoxon two-sample sensitivity.
- Rationale: Preserves unbiased inference if washout is insufficient.

#### 9.4 Diagnostics and robustness

Inspect residuals (fitted vs residuals, Q–Q) and influence (e.g., Cook's distance). If assumptions are violated, use robust (sandwich) SEs and confirm with a robust LMM or rank-based analysis; include the log-scale sensitivity if skewness persists.

## 10. Secondary analyses

# 10.1 Continuous change endpoints (SONG-Fatigue, STS-30, SF-12 PCS/MCS, labs, Kt/V)

LMM as in §9.1 (fixed: modality, period, sequence, centre; random: patient intercept; covariates per §8). Report adjusted mean difference (HDF – HD) with 95% CI.

## 10.2 Counts per period (hypotension, clotting)

Mixed-effects negative binomial model at patient–period level (fixed: modality, period, sequence, centre; random: patient intercept; offset = log[number of attended sessions]). If NB fails or over-dispersion negligible, use Poisson with robust SEs or a GEE sensitivity. Report rate ratio (HDF vs HD) with 95% CI.

#### 10.3 Safety (SAEs: deaths, hospitalizations)

Present exposure-adjusted incidence rates (EAIRs) per 100 patient-months by modality/period with 95% CIs. Optionally fit NB/Poisson models with offset = log(time on study in the period). No confirmatory testing.

#### 10.4 Subgroups (exploratory)

Pre-specified interactions of modality with: sex; age (85–89 vs ≥90); dialysis vintage (<2 vs ≥2 years); access type (AVF/AVG vs CVC); baseline fatigue tertiles; centre (e.g., enrolment size); convective volume tertiles (HDF only); dialysate buffer. Report interaction p-values (two-sided). Display forest plot. Interpretation exploratory (no multiplicity adjustment).

## 11. Missing data and exposure

- Windows: Require ≥2/3 session values to compute a window mean; otherwise missing.
- **Change endpoints:** Compute period-level change only when both Start and End windows are available; otherwise set period-level change to missing for that period.
- **Model-based handling:** Primary LMMs/NB models use all available patient–period records under MAR.
- Multiple imputation (robustness): Impute patient–period level changes using chained equations including modality, period, sequence, centre, baseline covariates, and auxiliary variables (e.g., session attendance, hospitalization indicator). Pool estimates via Rubin's rules.
- **Exposure adjustment:** For counts, include offsets as specified; sensitivity excluding periods with <27 attended sessions (~75% of planned 36 sessions).

## 12. Protocol deviations, adherence, and data cleaning

## 12.1 Major protocol deviations

- Incorrect eligibility after randomization (e.g., age <85; dialysis vintage <3 months).
- Washout not applied or <14 days at study start or between periods.
- Modality misclassification >20% of attended sessions in any period.
- Missing both Start or End windows for an endpoint in a period.
- Use of non-permitted procedures that materially affect endpoints.

#### 12.2 Adherence summaries

- Sessions attended per period; % sessions on allocated modality; mean convective volume (HDF); session duration; UF rate; temperature.
- Listings of crossovers and reasons (clinical need, access failure, etc.).

#### 12.3 Analysis by adherence

- Primary: ITT.
- Sensitivity: PP per above.
- Exploratory: As-treated using session-level exposure aggregated to period (e.g., ≥80% HDF vs ≥80% HD); IPTW sensitivity if meaningful confounding is suspected.

## 13. Interim analyses and data monitoring

No interim analyses or formal stopping rules are planned. Safety is monitored by the DSMB per protocol.

## 14. Software, reproducibility, and deliverables

- **Software:** Primary analyses in R (v4.3+).
- **Reproducibility:** Analysis code (R scripts, versions, sessionInfo) and TFL generation pipelines will be archived in the study repository with date/time stamps at database lock.
- **Deliverables:** TFLs in PDF/RTF; analyzable datasets and metadata (Analysis Data Model) retained per sponsor policy.

## 15. Tables, Figures, and Listings (TFLs) — overview

- Participant flow and disposition (CONSORT-style for crossover).
- Baseline characteristics by sequence and overall (Period-1 baseline).
- Treatment exposure/adherence per period and modality.
- **Primary endpoint:** Model summary ( $\beta_1$ , 95% CI, p), adjusted means by modality, diagnostic plots.
- Secondary endpoints: Change summaries and model outputs; counts with EAIRs.
- **Subgroups:** Forest plot of interaction effects.
- Safety: Listings of SAEs by modality/period; EAIR tables.